CLINICAL TRIAL: NCT01392131
Title: Study to Evaluate Safety and Therapeutic Efficacy of a Nutritional Supplement 'Oncoxin' in Patients With Hepatocellular Carcinoma
Brief Title: Safety and Efficacy of Oncoxin in Hepatocellular Carcinoma (HCC)
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Clinical Research Organization, Dhaka, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: OP1
Record Dates: First submitted 2011-07-07; First posted 2011-07-12 (Estimated); Last update posted 2012-12-12 (Estimated); Status verified 2012-12

CONDITIONS: Hepatocellular Carcinoma
Keywords: Oncoxin; Safety of Oncoxin; Therapeutic efficacy of Oncoxin; Improvement of quality of life with Oncoxin; Survival benefit with Oncoxin
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Viusid; Palliative Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oncoxin will be administered orally (Active Comparator): 20 patients will receive syrup Oncoxin 25 ml bd and capsule Oncoxin 1 cap bd for 24 weeks
  Interventions: Dietary Supplement: Oncoxin
- Supportive treatment (Active Comparator): 20 patients with hepatocellular carcinoma will receive supportive treatment only
  Interventions: Other: Supportive treatment

INTERVENTIONS:
Dietary Supplement: Oncoxin — 20 patients with hepatocellular carcinoma will receive syrup Oncoxin 25 ml bd and capsule Oncoxin 1 cap bd for 24 weeks
  Other Names: Viusid
  Arms: Oncoxin will be administered orally
Other: Supportive treatment — patients will receive only supportive treatment. No chemotherapy, radiotherapy, tumor ablation or surgery will be performed
  Arms: Supportive treatment

SUMMARY:
Oncoxin is safe and results in improved survival in patients with hepatocellular carcinoma

DETAILED DESCRIPTION:
To assess therapeutic efficacy and safety of Oncoxin in hepatocellular carcinoma

To see if there is reduction in serum alpha fetoprotein level in hepatocellular carcinoma patients after administration of Oncoxin

To see if there is reduction tumor size and or number in hepatocellular carcinoma patients after administration of Oncoxin

To see if there is improvement of quality of life in hepatocellular carcinoma patients after administration of Oncoxin

To see if there is improved survival in hepatocellular carcinoma patients after administration of oncoxin

ELIGIBILITY:
Inclusion Criteria:

* Patients with HCC irrespective of etiology, age, gender and status of underlying liver disease.
* Patients with HCC who are not suitable candidates for established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who have evidence of tumor metastasis
* Patients with HCC who are voluntarily unwilling to take established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC in whom all possible treatment options have been exhausted.

Exclusion Criteria:

* Patients with HCC who are suitable candidates for established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who have no evidence of tumor metastasis
* Patients with HCC who are willing to take established modalities of treatment i.e. surgery and/or chemotherapy.
* Patients with HCC who are voluntarily unwilling to be included in the trial

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2011-07; Primary Completion 2012-12 (Estimated); Study Completion 2013-07 (Estimated)

PRIMARY OUTCOMES:
Number of patients who have prolonged survival after receiving Oncoxin | 48 weeks
  To study the number of participants who have prolonged survival after receiving Oncoxin for 24 weeks.

SECONDARY OUTCOMES:
Reduction in serum alpha-fetoprotein level and decrease in tumor size | 48 weeks
  To see whether Oncoxin results in reduction in serum alpha-fetoprotein level and decrease in tumor size in hepatocellular carcinoma patients off treatment for 24 weeks, after receiving Oncoxin for 24 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Mamun A Mahtab, MSc MD FACG, Principal Investigator — Bangabandhu Sheikh Mujib Medical University, Dhaka, Bangladesh
Locations (1):
- Farabi General Hospital, Dhaka, Bangladesh